CLINICAL TRIAL: NCT01206556
Title: Duration of Human Papilloma Virus (HPV) Type-Specific Antibody After Administration of Quadrivalent HPV Vaccine (QHPV) to HIV-1 Infected Children Previously Enrolled in IMPAACT P1047
Brief Title: IMPAACT P1085: Human Papilloma Virus (HPV) Type-Specific Antibody
Acronym: HPV
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1085; U01AI068632 (NIH)
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Papilloma Virus, Human
Keywords: HUMAN PAPILLOMA VIRUS; HPV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is being done to evaluate how long the immune response from the Human Papilloma Virus (HPV) vaccine you / your child received persists. The immune response occurred after immunization and is what protects you/your child from HPV disease. You / your child received this vaccine as part of an earlier study (P1047). The vaccine is called Human Papillomavirus Vaccine (QHPV Vaccine, also known as GARDASIL®). The study will check to see if the protective effects (called "antibodies") produced by the vaccine have lasted, and for how long these effects will continue to last. You will not be given any medications or vaccines as part of this follow-up study.

DETAILED DESCRIPTION:
Genital Human Papilloma Virus (HPV) infection is the most common sexually transmitted infection (STI) in the United States and worldwide. Over 50% of sexually active adolescents will become infected with HPV. HPV infection is strongly associated with the development of anogenital dysplasias and invasive cancers. Because HPV is a STI, optimal prevention in women will depend on prevention in their partners as well. Males remain a significant reservoir of HPV and vaccinating them will be essential for rapidly preventing transmission of HPV in the community.

P1085 is a sub study of P1047, which investigated the safety and immunogenicity of Quadrivalent HPV (QHPV) in HIV-infected girls and boys, age 7 to <12 years of age. This study was a placebo-controlled trial that compared a recommended three dose schedule of QHPV in one study arm (Arm A) with an arm that received placebo (Arm B). P1047 has thus far demonstrated that QHPV can be safely administered to human immunodeficiency virus (HIV)-infected boys and girls and will stimulate seroconversion in more than 95% of vaccinees. However, these antibody levels were 30-50% lower than those achieved in children without HIV infection. Since levels of vaccine-induced antibodies decline with time after vaccination, it is uncertain if vaccine-induced immunity will be life-long. This concern is supported by some evidence that naturally acquired HPV-specific antibody might decline to a level that will permit re-infection. Comparative persistence data for HPV-specific antibody is available for 5-6 years after vaccination of almost 1000 children without HIV infection (manufacturer's data, unpublished), but there is no such information available from HIV-infected vaccinees.

We seek to determine the long-term durability and kinetics of the vaccine-induced HPV-type-specific antibody and CMI responses in HIV-infected children that were, and are being, immunized in P1047. These subjects are a unique cohort that will allow us to approach this specific clinical issue.

ELIGIBILITY:
Inclusion Criteria:

* Previous enrollment in P1047
* Completion of the P1047 scheduled vaccine doses for their designated arm.
* Parent or legal guardian able and willing to provide signed informed consent
* Subjects should be between 1 and 2 years following their last HPV vaccination.

Exclusion Criteria:

* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study.
* Administration of a globulin-containing product within 90 days prior to enrollment.
* Receipt of an additional dose of Merck HPV vaccine other than that administered for the P1047 study.
* Receipt of GSK HPV vaccine.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This will be limited to subjects who were enrolled into IMPAACT P1047 and who completed the scheduled vaccine doses for their designated arm.
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To determine the HPV-type specific antibody levels at 2, 3.5, and 5 years after completion of the QHPV vaccine schedule for each of the arms in P1047 | 208 weeks (4 Years)
  To determine the HPV-type specific antibody levels at 2, 3.5, and 5 years after completion of the QHPV vaccine schedule for each of the arms in P1047 and compare them to published levels of QHPV-induced antibody levels present in age-similar children IMPAACT P1085 without HIV infection at these time intervals after QHPV vaccination.

SECONDARY OUTCOMES:
Comparing the decline over the study interval in HPV type-specific antibody in subjects who received four doses of QHPV (Arm A) with those who received three doses of vaccine (Arm B) in P1047. | 4 years
  To compare the decline over the study interval in HPV type-specific antibody in subjects who received four doses of QHPV (Arm A) with those who received three doses of vaccine (Arm B) in P1047.
Determining the magnitude of HPV-specific antibody at different times after QHPV vaccination as a function of immune status (as defined by CD4 count and CD4 percent) and plasma HIV viral load. | 4 years
  To determine the magnitude of HPV-specific antibody at different times after QHPV vaccination as a function of immune status (as defined by CD4 count and CD4%) and plasma HIV viral load.
Determining the persistence of HPV-specific CMI at 2, 3.5, and 5 years after completion of the QHPV schedule for each of the arms in P1047. | 5 years after completion
  To determine the persistence of HPV-specific CMI at 2, 3.5, and 5 years after completion of the QHPV schedule for each of the arms in P1047.
Evaluating potential associations of HIV plasma RNA, lymphocyte immunophenotypes, HPV-specific memory B cell lymphocytes and HPV-specific CMI with the decay of anti-HPV antibody titers. | 4 years
  To evaluate potential associations of HIV plasma RNA, lymphocyte immunophenotypes, HPV-specific memory B cell lymphocytes and HPV-specific CMI with the decay of anti-HPV antibody titers.

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Levin, MD, Study Chair — University of Colorado, Denver
Locations (23):
- United States (22):
  - Miller Children's Hospital Long Beach (5093), Long Beach, California
  - USC/Los Angeles County Medical Center NICHD CRS (5048), Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CR (3601), Los Angeles, California
  - Univ of California, San Diego (4601), San Diego, California
  - Univ. of California San Francisco NICHD CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS (5052), Aurora, Colorado
  - Children's National Med. Ctr. Washington DC NICHD CRS (5015), Washington D.C., District of Columbia
  - South Florida CDC Ft. Lauderdale NICHD CRS (5055), Fort Lauderdale, Florida
  - Univ of Miami Pediatric/Perinatal HIV/AIDS (4201), Miami, Florida
  - Rush University Cook County Hospital NICHD CRS (5083), Chicago, Illinois
  - Chicago Children's CRS (4001), Chicago, Illinois
  - Children's Hospital of Boston (5009), Boston, Massachusetts
  - Boston Medical Center Ped. HIV Program NICHD CRS (5011), Boston, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS (7301), Worcester, Massachusetts
  - Wayne State University/Children's Hospital of Michigan NICHD CRS (5041), Detroit, Michigan
  - New Jersey Medical School (NJ) (2802), Newark, New Jersey
  - New York University NY (5012), New York, New York
  - Strong Memorial Hospital, University of Rochester NICHD CRS (5057), Rochester, New York
  - SUNY Stony Brook (5040), Stony Brook, New York
  - Bronx-Lebanon Hospital (6901), The Bronx, New York
  - Jacobi Medical Center Bronx (5013), The Bronx, New York
  - Texas Children's Hosp / Baylor Univ (3801), Houston, Texas
- San Juan City Hosp. PR NICHD CRS (5031), San Juan, Puerto Rico

REFERENCES:
- [Derived] Levin MJ, Huang S, Moscicki AB, Song LY, Read JS, Meyer WA, Saah AJ, Richardson K, Weinberg A; IMPAACT P1085 Protocol Team. Four-year persistence of type-specific immunity after quadrivalent human papillomavirus vaccination in HIV-infected children: Effect of a fourth dose of vaccine. Vaccine. 2017 Mar 23;35(13):1712-1720. doi: 10.1016/j.vaccine.2017.02.021. Epub 2017 Feb 24. PMID 28238631
- See also: IMPAACT Network Web Site — http://impaactgroup.org